CLINICAL TRIAL: NCT06581185
Title: Headache Long Term Follow-up in Patients Who Suffered From PTCS During Their Childhood
Brief Title: Pseudotumor Cerebri Headache Ten Years Outcome
Status: Enrolling by invitation | Type: Observational
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: BNAI ZION MEDICAL CENTER
Record Dates: First submitted 2024-08-27; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Pseudotumor Cerebri
Keywords: Headache; outcome
MeSH Terms: conditions — Pseudotumor Cerebri; Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Research: Patients who were diagnosed with PTC as children

SUMMARY:
Telephone interview on patient who suffered from PTC ten years ago regarding their headache status

DETAILED DESCRIPTION:
The study will followup using existing medical data from patients previously diagnosed with Pseudotumor cerebri (PTC) using a telephone contact with patients diagnosed more than 10 years ago. After obtaining verbal consent, conducted interviews to collect information on their headaches and quality of life. Data related to PTC was be obtained from medical records. Demographic information was be collected using a questionnaire, the HIT-6 questionnaire will assess headache severity, and a quality of life questionnaire was be used.

ELIGIBILITY:
Inclusion Criteria:

Patients who were diagnosed with PTC as children

-

Exclusion Criteria:

Patients has other headache types other than PTC

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults who were diagnosed with Ptc at their childhood .
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
headache outcome HIT-6 | 5-10 years
  How many patients will suffer from headache after recovery from PTC measured by HIT 6 questionnaire

SECONDARY OUTCOMES:
Quality of life (QOL) | 5-10 years
  Is the QOL of patients recovering from PTS related to their headache measured by WHO QOL questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: jacob Genizi, Principal Investigator — Bnai Zion Medical Center
Locations (1):
- Bani Zion, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Smith JL. Whence pseudotumor cerebri? J Clin Neuroophthalmol. 1985 Mar;5(1):55-6. No abstract available. PMID 3156890
- [Result] Kesler A, Bassan H. Pseudotumor cerebri - idiopathic intracranial hypertension in the pediatric population. Pediatr Endocrinol Rev. 2006 Jun;3(4):387-92. PMID 16816807
- [Result] Buchheit WA, Burton C, Haag B, Shaw D. Papilledema and idiopathic intracranial hypertension. N Engl J Med. 1969 Apr 24;280(17):938-42. doi: 10.1056/NEJM196904242801707. No abstract available. PMID 5775633
- [Result] Friedman DI, Jacobson DM. Diagnostic criteria for idiopathic intracranial hypertension. Neurology. 2002 Nov 26;59(10):1492-5. doi: 10.1212/01.wnl.0000029570.69134.1b. PMID 12455560
- [Result] Baker RS, Baumann RJ, Buncic JR. Idiopathic intracranial hypertension (pseudotumor cerebri) in pediatric patients. Pediatr Neurol. 1989 Jan-Feb;5(1):5-11. doi: 10.1016/0887-8994(89)90002-7. PMID 2653341
- [Result] Couch R, Camfield PR, Tibbles JA. The changing picture of pseudotumor cerebri in children. Can J Neurol Sci. 1985 Feb;12(1):48-50. doi: 10.1017/s0317167100046588. PMID 3978475
- [Result] Dhiravibulya K, Ouvrier R, Johnston I, Procopis P, Antony J. Benign intracranial hypertension in childhood: a review of 23 patients. J Paediatr Child Health. 1991 Oct;27(5):304-7. doi: 10.1111/j.1440-1754.1991.tb02544.x. PMID 1931224

DOCUMENTS (1):
  • Study Protocol (2024-07-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT06581185/Prot_000.pdf